CLINICAL TRIAL: NCT02516410
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of VX-661 in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Heterozygous for the F508del-CFTR Mutation and With a Second CFTR Mutation That Is Not Likely to Respond to VX-661 and/or Ivacaftor Therapy (F508del/NR)
Brief Title: A Study to Evaluate the Efficacy and Safety of VX-661 in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Heterozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX14-661-107; 2014-004787-37 (EudraCT Number)
Record Dates: First submitted 2015-07-28; First posted 2015-08-05 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VX-661/IVA (Experimental): VX-661 100 milligram (mg) plus IVA 150 mg fixed dose combination (FDC) tablet administered orally in the morning and IVA 150 mg film-coated tablet administered orally in the evening up to Week 12.
  Interventions: Drug: VX-661 plus ivacaftor combination; Drug: Ivacaftor
- Placebo (Placebo Comparator): Placebo matched to VX-661 plus IVA FDC tablet administered orally in the morning and placebo matched to IVA film-coated tablet administered orally in the evening up to Week 12.
  Interventions: Drug: Placebo (matched to VX-661 plus ivacaftor combination); Drug: Placebo (matched to ivacaftor)

INTERVENTIONS:
Drug: VX-661 plus ivacaftor combination
  Arms: VX-661/IVA
Drug: Ivacaftor
  Other Names: IVA; VX-770
  Arms: VX-661/IVA
Drug: Placebo (matched to VX-661 plus ivacaftor combination)
  Arms: Placebo
Drug: Placebo (matched to ivacaftor)
  Arms: Placebo

SUMMARY:
Study to evaluate the efficacy of VX-661 in combination with ivacaftor (IVA, VX-770) through Week 12 in participants with cystic fibrosis (CF) who are heterozygous for the F508del mutation on the CF transmembrane conductance regulator (CFTR) gene and with a second CFTR mutation that is not likely to respond to VX-661 and/or IVA therapy (F508del/not responsive [NR]).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF defined as a sweat chloride value greater than or equal to (>=)60 millimole per liter (mmol/L) by quantitative pilocarpine iontophoresis.
* Heterozygous for the F508del-CFTR mutation and with a second CFTR mutation that is not likely to respond to VX-661 and/or ivacaftor therapy, genotype to be confirmed via assessment at the Screening Visit.
* Forced Expiratory Volume in 1 Second (FEV1) >=40 percent (%) and less than or equal to (<=)90% of predicted normal for age, sex, and height at Screening Visit.

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 28 days before Day 1 (first dose of study drug).
* History of solid organ or hematological transplantation.
* Ongoing or prior participation in an investigational drug study or use of commercially available CFTR modulator within 30 days of screening.
* Pregnant or nursing females.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (22):
  - Birmingham, Alabama
  - La Jolla, California
  - Los Angeles, California
  - Denver, Colorado
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Cincinnati, Ohio
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Australia (5):
  - Brisban, Queensland
  - Chermside
  - Herston
  - Innsbruck
  - Westmead
- Austria (3):
  - Graz
  - Innsbruck
  - Salzburg
- Canada (2):
  - Vancouver, British Columbia
  - Montreal
- France (3):
  - Bron
  - Montpellier
  - Paris
- Israel (4):
  - Haifa
  - Hashomer
  - Jerusalem
  - Petah Tikva
- Spain (2):
  - Barcelona
  - Valencia

REFERENCES:
- [Derived] Munck A, Kerem E, Ellemunter H, Campbell D, Wang LT, Ahluwalia N, Owen CA, Wainwright C. Tezacaftor/ivacaftor in people with cystic fibrosis heterozygous for minimal function CFTR mutations. J Cyst Fibros. 2020 Nov;19(6):962-968. doi: 10.1016/j.jcf.2020.04.015. Epub 2020 Jun 13. PMID 32546431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 38 sites in 7 countries.
Pre-assignment Details: A total of 168 participants were randomized and treated in the study.
Groups:
- Placebo: Placebo matched to VX-661 plus Ivacaftor (IVA, VX-770) fixed dose combination (FDC) tablet administered orally in the morning and placebo matched to IVA film-coated tablet administered orally in the evening up to Week 12.
- VX-661/IVA: VX-661 100 milligram (mg) plus IVA 150 mg FDC tablet administered orally in the morning and IVA 150 mg film-coated tablet administered orally in the evening up to Week 12.
Period: Overall Study
Arm/Group | Placebo | VX-661/IVA
Started | 85 | 83
Completed | 85 | 81
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- VX-661/IVA: VX-661 100 mg plus IVA 150 mg FDC tablet administered orally in the morning and IVA 150 mg film-coated tablet administered orally in the evening up to Week 12.
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-661/IVA | Total
Number analyzed (Participants) | 85 | 83 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (8.8) | 26.2 (9.6) | 26.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 81
  Male | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 12
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years.
Time Frame: Baseline, Through Week 12
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug. Here 'Number of participants analysed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of predicted FEV1
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 82
Percentage of predicted FEV1 | -0.1 (0.6) | 1 (0.6)
Statistical Analysis 1: Comparison: Placebo vs VX-661/IVA; Test type: Superiority; p = 0.1176, Mixed-effect repeated measure (MMRM); Least squares (LS) mean difference = 1.2, 95% CI 2-sided [-0.3 to 2.6]

2. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 12
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Through Week 12
Population: FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 83
Units on a scale | 3.8 [1.1 to 6.4] | 5.9 [3.2 to 8.5]

3. Secondary Outcome: Number of Pulmonary Exacerbation Events
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. The number of events were reported.
Time Frame: Baseline through Week 12
Population: FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Pulmonary exacerbation events
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 83
Pulmonary exacerbation events | 23 | 22

4. Secondary Outcome: Number of Pulmonary Exacerbation Events Per Year
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Total number of days on study is equal to the Week 12 date or the last dose date (whichever occurs last) minus first dose date plus 1. The total number of years (48 weeks) on study is equal to the total number of days on study divided by 336. Pulmonary exacerbation events per year (48 weeks) are reported.
Time Frame: Baseline through Week 12
Population: FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Pulmonary exacerbation events per year
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 83
Pulmonary exacerbation events per year | 0.98 | 0.97

5. Secondary Outcome: Absolute Change From Baseline in Body Mass Index (BMI) at Week 12
Description: BMI was defined as weight in kilogram (kg) divided by height*height in square meter (m^2).
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants who received at least 1 dose of study drug. Here 'Number of participants analysed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kg/m^2
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 82
Kg/m^2 | 0.22 [0.07 to 0.36] | 0.14 [-0.01 to 0.28]

6. Secondary Outcome: Relative Change From Baseline in Percent Predicted FEV1 Through Week 12
Description: as for outcome 1
Time Frame: Baseline, Through Week 12
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 82
Percent Change | 0.1 [-2.1 to 2.3] | 2.1 [-0.1 to 4.3]

7. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride Through Week 12
Description: Sweat samples were collected using an approved collection device.
Time Frame: Baseline, Through Week 12
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimole per liter (mmol/L)
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 84 | 79
Millimole per liter (mmol/L) | -1.2 [-3.1 to 0.7] | -4.7 [-6.6 to -2.8]

8. Secondary Outcome: Number of Participants With at Least One Pulmonary Exacerbation Through Week 12
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Time-to-first pulmonary exacerbation was planned to be estimated using Kaplan-Meier (KM) estimates. However, due to less than 50% of events, time-to-first event data was not estimated. Instead, number of participants with at least one pulmonary exacerbation event were collected and are reported.
Time Frame: Baseline through Week 12
Population: FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 83
Participants | 21 | 19

9. Secondary Outcome: Absolute Change From Baseline in BMI Z-score at Week 12 (in Participants Less Than [<] 20 Years Old at the Time of Screening)
Description: Z-score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard and how unusual the measurement is, with range from infinity to +infinity; where 0: same mean, >0: a greater mean, and <0: a lesser mean than the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age Z-score (BMI z-score). BMI-for-age z-score was calculated by using centers for disease control and prevention (CDC) growth charts for the paediatric population.
Time Frame: Baseline, Week 12
Population: Analysis population included all randomized participants who received at least 1 dose of study drug and were <20 years of age at the time of screening.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 22 | 25
Z-score | 0.07 [-0.05 to 0.19] | 0.02 [-0.09 to 0.13]

10. Secondary Outcome: Absolute Change From Baseline in Body Weight at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms (kg)
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 82
Kilograms (kg) | 0.7 [0.3 to 1.1] | 0.6 [0.2 to 1.0]

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Any AE that increased in severity or newly developed at or after initial dosing of study drug to Week 16 was considered treatment-emergent.
Time Frame: Baseline up to Week 16
Population: Safety Set included all participants who received at least 1 dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 85 | 83
Participants
  Participants with any AEs | 68 | 64
  Participants with any SAEs | 14 | 11

12. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of VX-661, VX-661 Metabolite (M1 VX-661), Ivacaftor (IVA) and IVA Metabolite (M1-IVA)
Description: This outcome was not planned to be assessed in Placebo arm.
Time Frame: Pre-morning dose on Week 2, Week 4, Week 8 and Week 12
Population: Pharmacokinetic (PK) set included all randomized participants who received any amount of study drug and had a PK assessment. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | VX-661/IVA
Number analyzed (Participants) | 82
nanogram per milliliter (ng/mL)
  Week 2: VX-661: number analyzed (Participants) | 80
  Week 2: VX-661 | 1880 (1230)
  Week 2: M1 VX-661: number analyzed (Participants) | 80
  Week 2: M1 VX-661 | 4600 (1430)
  Week 2: IVA: number analyzed (Participants) | 79
  Week 2: IVA | 831 (607)
  Week 2: M1-IVA: number analyzed (Participants) | 79
  Week 2: M1-IVA | 1580 (879)
  Week 4: VX-661 | 1780 (1010)
  Week 4: M1 VX-661 | 4420 (1340)
  Week 4: IVA | 770 (596)
  Week 4: M1-IVA | 1500 (898)
  Week 8: VX-661: number analyzed (Participants) | 80
  Week 8: VX-661 | 1920 (2170)
  Week 8: M1 VX-661: number analyzed (Participants) | 80
  Week 8: M1 VX-661 | 4330 (1980)
  Week 8: IVA: number analyzed (Participants) | 81
  Week 8: IVA | 747 (745)
  Week 8: M1-IVA: number analyzed (Participants) | 81
  Week 8: M1-IVA | 1370 (1070)
  Week 12: VX-661: number analyzed (Participants) | 81
  Week 12: VX-661 | 1700 (1220)
  Week 12: M1 VX-661: number analyzed (Participants) | 81
  Week 12: M1 VX-661 | 4290 (1730)
  Week 12: IVA: number analyzed (Participants) | 81
  Week 12: IVA | 776 (690)
  Week 12: M1-IVA: number analyzed (Participants) | 81
  Week 12: M1-IVA | 1620 (1160)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Arm/Group | Placebo | VX-661/IVA
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/83
Serious Adverse Events (participants affected / at risk) | 14/85 | 11/83
Other Adverse Events (participants affected / at risk) | 63/85 | 62/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | VX-661/IVA (N=83)
Pulmonary function test decreased (Investigations) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 12 | 6
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | VX-661/IVA (N=83)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 19
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Headache (Nervous system disorders) | 7 | 5
Fatigue (General disorders) | 4 | 10
Pyrexia (General disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 6 | 6
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 15 | 17
Nasopharyngitis (Infections and infestations) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: PI is free to publish results of the study after (1)first multi-center publication, (2)if sponsor elects not to publish the results, or (3)18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications